CLINICAL TRIAL: NCT07386743
Title: A Multicenter, Randomized, Double-blinded, Parallel, Positive-controlled, Phase III Comparative Study to Evaluate GS101 Injection Versus Dupixent® in Participants With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Phase III Study of GS101 Injection to Dupixent®
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Genscend Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS101-03
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — GS 101; dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS101 injection (Experimental)
  Interventions: Drug: GS101 injection
- Dupixent® (Active Comparator)
  Interventions: Drug: DUPIXENT®

INTERVENTIONS:
Drug: GS101 injection — 300mg/2.0mL; an initial dose of 600 mg (two 300 mg injections), followed by 300 mg given every other week (Q2W);subcutaneous injection
  Arms: GS101 injection
Drug: DUPIXENT® — 300mg/2.0mL; an initial dose of 600 mg (two 300 mg injections), followed by 300 mg given every other week (Q2W); subcutaneous injection
  Arms: Dupixent®

SUMMARY:
This is a a multicenter, randomized, double-blinded, parallel, positive-controlled, Phase III comparative study to evaluate GS101 Injection versus Dupixent® in participants with moderate-to-severe atopic dermatitis. A total of 572 subjects are planned to be included and randomized at a ratio of 1:1 to receive GS101 injection or Dupixent®

ELIGIBILITY:
Inclusion Criteria:

* Subjects, male or female, between the ages of 18 and 75 years (inclusive)
* At the time of screening, the diagnosis of atopic dermatitis (AD) meets the Hanifin-Rajka criteria, with a disease history for at least 1 year prior to screening
* During the screening period and at baseline, patients with moderate-to-severe atopic dermatitis, defined as meeting all of the following 3 criteria concurrently: a. IGA score ≥ 3; b. EASI score ≥ 16; c. BSA ≥ 10%.

Exclusion Criteria:

* Hypersensitivity or known allergy to the investigational product(s) or any of their excipients
* Treatment with any investigational drug, medical device, or other biologic agent within 8 weeks prior to randomization or within 5 half-lives (if the half-life is known), whichever is longer
* Receipt of any live or live-attenuated vaccine within 3 months prior to randomization, or planned receipt of such vaccines during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving EASI-75 at week 16 | 16 weeks
  EASI-75

SECONDARY OUTCOMES:
Proportion of patients achieving EASI-75 | Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, and 52
  Proportion of patients achieving EASI-50 at Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, and 52
Proportion of patients achieving EASI-50 | Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, and 52
  Proportion of patients achieving EASI-50 at Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, and 52
Proportion of patients achieving EASI-90 | Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, and 52
  Proportion of patients achieving EASI-90 at Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, and 52

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China